CLINICAL TRIAL: NCT02328937
Title: Daily Wear Central Corneal Swelling With Etafilcon A and 2 Silicone Hydrogel Materials
Brief Title: Central Corneal Swelling With Silicone Hydrogel Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR-5550
Record Dates: First submitted 2014-12-03; First posted 2014-12-31 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-12

CONDITIONS: Corneal Swelling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- etafilcon A/lotrafilcon B/comfilcon A (Active Comparator): Subjects that were randomized to receive the etafilcon A lens 1st, the lotrafilcon B lens 2nd and the comfilcon A lens 3rd.
  Interventions: Device: etafilcon A; Device: lotrafilcon B; Device: comfilcon A
- etafilcon A/comfilcon A/lotrafilcon B (Active Comparator): Subjects that were randomized to receive the etafilcon A lens 1st, the comfilcon A lens 2nd and the lotrafilcon B lens 3rd.
  Interventions: Device: etafilcon A; Device: lotrafilcon B; Device: comfilcon A
- comfilcon A/etafilcon A/lotrafilcon B (Active Comparator): Subjects that were randomized to receive the comfilcon A lens 1st, the etafilcon A lens 2nd and the lotrafilcon B lens 3rd.
  Interventions: Device: etafilcon A; Device: lotrafilcon B; Device: comfilcon A
- comfilcon A/lotrafilcon B/etafilcon A (Active Comparator): Subjects that were randomized to receive the comfilcon A lens 1st, the lotrafilcon B lens 2nd and the etafilcon A lens 3rd.
  Interventions: Device: etafilcon A; Device: lotrafilcon B; Device: comfilcon A
- lotrafilcon B/etafilcon A/comfilcon A (Active Comparator): Subjects that were randomized to receive the lotrafilcon B lens 1st, the etafilcon A lens 2nd and the comfilcon A lens 3rd.
  Interventions: Device: etafilcon A; Device: lotrafilcon B; Device: comfilcon A
- lotrafilcon B/comfilcon A/etafilcon A (Active Comparator): Subjects that were randomized to receive the lotrafilcon B lens 1st, the comfilcon A lens 2nd and the etafilcon A lens 3rd.
  Interventions: Device: etafilcon A; Device: lotrafilcon B; Device: comfilcon A

INTERVENTIONS:
Device: etafilcon A — spherical hydrophilic soft contact lens worn in a daily wear modality
  Other Names: Investigational Soft Contact Lens -
Device: lotrafilcon B
Device: comfilcon A

SUMMARY:
This is a prospective, single site, unmasked, cross-over study with three silicone hydrogel contact lenses comparing central corneal swelling.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be at leat 18 years old or older and no greater than 65 years old. Children younger than18 will likely no be able to come back and forth to the clinic during the typical work week as outlined in the above (due to school schedules) and thus not be able to adhere to the protocol.
2. The participant must be a current soft contact lens wearer who routinely wears lenses at least 6-8 hours per day and at least 4 days per week for at least the past 3 months.
3. Refraction suitable for spherical soft contact lens powers between -1.00 and -6.00 D the participant must be correctable to 20/30 or better at distance with both eyes with dispensed contact lenses.
4. The participant must be free of any active anterior segment disorders that would preclude safe contact lens wear. Active anterior segment disorders and evidence of central microbial keratitis are not allowed. However, evidence of past CLPU will be allowed so long as no more than 3 such scars are detected bilaterally. Evidence of more than 3 CLPU-like scars places excessive risk on the participant for subsequent CIE.
5. The participant must be correctable to 20/25 or better in each eye with spectacles. Amblyopia will be excluded.
6. Flat and steep corneal curvatures from keratometry readings must be between 39.00 and 48.50 D, respectively. Corneal curvatures outside this range may be indicative of a disease state, and the participants are not expected to comfortably wear the study lenses.
7. The participant must own or agree to purchase a pair of spectacles that can be worn when lenses are removed, during the washout periods, or in case of ocular discomfort or emergency.

Exclusion Criteria:

1. The participant has worn rigid gas permeable contact lenses within the last 30 days or PMMA lenses within the past 12 months. These lenses can transiently alter the corneal shape and influence the fitting of soft contact lenses or alter endothelial cell morphology.
2. The participant has an immunocompromising disease or any other systemic disease that in the investigator's opinion will affect ocular health or increase risk during daily contact lens wear.
3. The participant is taking any medication that in the investigator's opinion will affect ocular physiology or study participation.
4. The participant has an ocular disease or condition such as aphakia, clinically significant corneal dystrophies, corneal edema, external ocular infection, iritis, or had any anterior segment surgery.
5. The participant is taking any ocular medications. If a participant was previous taking any ocular medications, the medications must have been discontinued at least 2 weeks prior to enrollment.
6. The participant must have less than or equal to grade 2 on any of the slit lamp observations of: upper tarsal papilla, corneal staining, corneal neovascularization, conjunctival injection, and lid erythema or scales.
7. The participant is currently pregnant or lactating. Participant who become pregnant during the study will be discontinued.
8. An employee or member of the UHCMC Eye Institute or a family member of any study personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 subjects were enrolled in this study. Of the enrolled subjects 3 did not meet the eligibility criteria and 38 subjects were dispensed a study lens. Of the dispensed subjects 2 were discontinued while 36 completed all study visits.
Groups:
- Etafilcon A/Lotrafilcon B/Comfilcon A: Subjects randomized to this sequence received etafilcon A during the 1st period, then received lotrafilcon B during the 2nd period, and then received comfilcon A during the last period.
- Etafilcon A/Comfilcon A/Lotrafilcon B: Subjects randomized to this sequence received etafilcon A during the 1st period, then received comfilcon A during the 2nd period, and then received lotrafilcon B during the last period.
- Lotrafilcon B/Etafilcon A/Comfilcon A: Subjects randomized to this sequence received lotrafilcon B during the 1st period, then received etafilcon A during the 2nd period, and then received comfilcon A during the last period.
- Lotrafilcon B/Comfilcon A/Etafilcon A: Subjects randomized to this sequence received lotrafilcon B during the 1st period, then received comfilcon A during the 2nd period, and then received etafilcon A during the last period.
- Comfilcon A/Etafilcon A/Lotrafilcon B: Subjects randomized to this sequence received comfilcon A during the 1st period, then received etafilcon A during the 2nd period, and then received lotrafilcon B during the last period.
- Comfilcon A/Lotrafilcon B/Etafilcon A: Subjects randomized to this sequence received comfilcon A during the 1st period, then received lotrafilcon B during the 2nd period, and then received etafilcon A during the last period.
Period: Period 1
Arm/Group | Etafilcon A/Lotrafilcon B/Comfilcon A | Etafilcon A/Comfilcon A/Lotrafilcon B | Lotrafilcon B/Etafilcon A/Comfilcon A | Lotrafilcon B/Comfilcon A/Etafilcon A | Comfilcon A/Etafilcon A/Lotrafilcon B | Comfilcon A/Lotrafilcon B/Etafilcon A
Started | 7 | 6 | 7 | 6 | 6 | 6
Completed | 7 | 6 | 7 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Etafilcon A/Lotrafilcon B/Comfilcon A | Etafilcon A/Comfilcon A/Lotrafilcon B | Lotrafilcon B/Etafilcon A/Comfilcon A | Lotrafilcon B/Comfilcon A/Etafilcon A | Comfilcon A/Etafilcon A/Lotrafilcon B | Comfilcon A/Lotrafilcon B/Etafilcon A
Started | 7 | 6 | 7 | 5 | 6 | 6
Completed | 7 | 6 | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | Etafilcon A/Lotrafilcon B/Comfilcon A | Etafilcon A/Comfilcon A/Lotrafilcon B | Lotrafilcon B/Etafilcon A/Comfilcon A | Lotrafilcon B/Comfilcon A/Etafilcon A | Comfilcon A/Etafilcon A/Lotrafilcon B | Comfilcon A/Lotrafilcon B/Etafilcon A
Started | 7 | 6 | 6 | 5 | 6 | 6
Completed | 7 | 6 | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Overall: All subjects that were dispensed at least one study lens.
Arm/Group | Overall
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 9
  Black or African American | 10
  White | 19
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Central Corneal Swelling
Description: Corneal swelling measurements were taken in the right eye during slit lamp evaluations, 6-8 hours post lens insertion. The average corneal swelling per lens was reported.
Time Frame: 6-8 Hours Post lens insertion
Population: All subjects that were dispensed at least one study lens throughout the duration of the study.
Measure: Mean (Standard Deviation); unit: um
Groups:
- Etafilcon A: Subjects that wore the etafilcon A lens during any of the 3 period over the course of this study.
- Lotrafilcon B: Subjects that wore the lotrafilcon B lens during any of the 3 period over the course of this study.
- Comfilcon A: Subjects that wore the comfilcon A lens during any of the 3 period over the course of this study.
Arm/Group | Etafilcon A | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 37 | 38 | 36
um | 542.2 (31.28) | 542.4 (30.69) | 544.3 (28.30)

2. Secondary Outcome: Limbal Redness
Description: Limbal redness was assessed in both eyes using a slit lamp, 6-8 hours post lens insertion. Redness was assessed in 4 regions of the eye (nasal, temporal, inferior and superior) and was graded with a 5-point scale (i.e. Grade 0= None, Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). For each region (nasal, temporal, inferior and superior) the average grade was calculated by lens. The Total Grade was then calculated by summing all the average grade for each region. The regional average grade ranges from 0 to 4. The total Grade ranges from 0 to 16.
Time Frame: 6-8 hours post lens insertion
Population: All subjects that were dispensed at least one study lens throughout the duration of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etafilcon A | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 37 | 38 | 36
units on a scale | 6.46 (1.233) | 6.24 (1.177) | 6.14 (0.977)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration. Approximately 1-week per subject
Arm/Group | Etafilcon A | Lotrafilcon B | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days